CLINICAL TRIAL: NCT03041974
Title: Cell-derived Microparticles in Red Blood Cell (RBC) Concentrates, and Their Potential Impact on Outcomes of Transfused Patients in Critical Care: a Prospective Multicentre National Cohort Study of Patients Included in the ABLE Trial
Brief Title: Impact of Microparticles in Blood on Transfused Patient Outcomes
Acronym: IMIB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: IMIB PHRC 2013
Record Dates: First submitted 2016-09-12; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Critical Care
Keywords: Red Blood Cell Transfusion; Cell-Derived Microparticles
MeSH Terms: interventions — Erythrocyte Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transfused critical care patients: Patients included in the Age of BLood Evaluation (ABLE) trial in either arms and included in a French center.
  Interventions: Procedure: Red Blood Cell transfusion; Procedure: Microparticles quantification

INTERVENTIONS:
Procedure: Red Blood Cell transfusion
Procedure: Microparticles quantification — Flow cytometric quantification of microparticles in transfused blood

SUMMARY:
During storage, red blood cells (RBCs) undergo changes collectively termed "Storage lesions". these changes may have an impact of the outcomes of transfused patients. One of these changes is the release of microparticles by RBCs and other blood cells types. The aim of the study is to (1) quantify red cell- and platelet-derived microparticles in RBC concentrates, and (2) evaluate the impact of transfused microparticles (MPs) on survival and post-transfusion complications in critical care patients participating in the ABLE trial (ISRCTN44878718).

DETAILED DESCRIPTION:
During conservation of red blood cell concentrates, red blood cells (RBCs) undergo biochemical and morphological changes that have been well described, and are collectively termed " storage lesions ". The exact effects of these lesions in terms of beneficial or deleterious implications in the recipient remain to be elucidated. However, several retrospective studies in targeted populations suggest that an increase in the duration of RBC conservation could lead to an increase in morbidity and mortality in transfused patients. The multicenter, prospective trial ABLE (Age of Blood Evaluation, ISRCTN44878718) aimed to evaluate in a randomised clinical trial, the impact of the age of transfused RBC concentrates on several outcomes in critical care patients.

Among the modifications that RBCs undergo during storage, the generation of microparticles from red blood cellsRBCs or residual platelets present in the blood concentrate has never been evaluated in a prospective clinical study. It has been reported that the number of red cell-derived microparticles (RMPs) present in stored blood increases with storage duration. In vivo, microparticles MPs appear to be increasingly involved in disease processes, notably due to their pro-inflammatory and pro-coagulant effects. Furthermore, it has been shown that the antigens of the Rhesus group are expressed on the RBC derived microparticles, and the investigative team has shown that microparticles derived from elsewhere (endothelial cells) are capable of activating cells which are important in the induction of immune responses (dendritic cells). Thus, transfusing red blood cell derived microparticles could participate in post-transfusional alloimmunization which may also be evaluated in this study.

The aim of the IMIB study is to (1) quantify red cell- and platelet-derived microparticles MPs in RBC concentrates, and (2) evaluate the impact of the quantity of transfused microparticles (MPs) on survival and several outcomes in the patients enrolled in the ABLE trial in France.

Other aims are to investigate the relationship between the number of microparticles in RBC units and (1) the age of RBC, (2) donors characteristics, (3) the procedures used to prepare the blood products (to define a potential new "lesion storage" marker).

ELIGIBILITY:
Inclusion Criteria are those of the ABLE trial: patients who

* Have had a request for a first red cell unit transfusion in the Intensive Care Unit (ICU), and
* Have an anticipated length of invasive and/or non-invasive continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BIPAP) mechanical ventilation of at least 48 hours once enrolled, as estimated by the attending physician

Exclusion Criteria:

* less than 18 years of age
* previously enrolled in the ABLE study
* has already been transfused with red cells during the current hospitalisation
* has an obvious terminal illness documented in the medical record with a life expectancy of less than 3 months
* has undergone routine cardiac surgical care
* decision to withdraw/withhold some critical care had been made
* brain dead
* no red cells with a storage time of 7 days or less available in the blood bank that cannot be transported from the blood supplier
* Who require more than 1 unit of uncross-matched red cells
* With a known objection to blood transfusions
* With autologous blood donations
* Who pose difficulties in securing blood products (rare blood groups), and who are difficult to match

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are the patients enrolled, by french centers, in either arms of the ABLE trial.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 90 days

SECONDARY OUTCOMES:
All cause mortality | 28 days, 6 months
Multi organ dysfunction score | 6 months
Nosocomial infection | 6 months
  including Nosocomial pneumonia, Deep tissue infections (e.g. peritonitis, mediastinitis), Bacteraemia from organisms not considered normal skin flora and judged important enough to treat by the attending team, as measured while in the ICU

OTHER OUTCOMES:
Intensive care and Hospital duration of stay | 6 months
Length of time requiring respiratory, haemodynamic and renal support | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francine Garnache-Ottou, PharmD, PhD, Principal Investigator — Etablissement Français du Sang, Besançon

IPD SHARING:
Plan to Share IPD: No